CLINICAL TRIAL: NCT06384651
Title: Intraosseous vs. Intravenous Vancomycin Administration in Total Ankle Arthroplasty
Acronym: IOTAA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jason S. Ahuero, Orthopedic Surgeon, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00037789
Record Dates: First submitted 2024-04-02; First posted 2024-04-25 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Infections; Ankle Arthritis
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, single-blinded, controlled trial. 20 patients in each treatment arm: 20 patients will be given IV vancomycin, 20 patients will be given IO vancomycin
Who Masked: Participant, Outcomes Assessor
Masking Description: single blind patient is blinded. Surgeon is not blinded. Lab technician measuring tissue concentrations are blinded. Research coordinator is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Vancomycin (Active Comparator): Patients will receive the orthopedic surgeon's standard of care pre-operative antibiotic regimen for TAA patients. This includes IV antibiotics (typically ancef or cefepime and vancomycin) will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg generally 1000-1750mg in 500mL normal saline (NS))
  Interventions: Drug: Intravenous Vancomycin
- Intraosseous Vancomycin (Experimental): IV antibiotics per physician's standard of care: Typically ancef or cefepime is started in pre-op within 1 hour of incision. IV Vancomycin will not be given preoperatively in this group.
  IO vancomycin is administered in the OR after sterile prep and draping has occurred (500mg in 100-150mL NS).
  IO Injection will take place into the medial malleolus.
  Interventions: Drug: Intraosseous Vancomycin Injection

INTERVENTIONS:
Drug: Intraosseous Vancomycin Injection — * IO vancomycin is administered in the OR after sterile prep and draping has occurred (500mg in 100-150mL NS).
  * IO Injection will take place into the medial malleolus.
  Arms: Intraosseous Vancomycin
Drug: Intravenous Vancomycin — • Patients will receive the orthopedic surgeon's standard of care pre-operative antibiotic regimen for TAA patients. This includes IV antibiotics (typically ancef or cefepime and vancomycin) will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg generally 1000-1750mg in 500mL normal saline (NS))
  Arms: Intravenous Vancomycin

SUMMARY:
The purpose of this study is to compare two different antibiotic regimens and techniques during total ankle arthroplasty (TAA).

Primary Objective: Comparable levels of vancomycin will be found in bone, soft tissue, and systemic samples between patient groups.

Secondary Objective: Compare 30 day and 90 day post-operative complication rates (infection) between the control (standard IV administration of vancomycin) vs the interventional group (intraosseous administration of vancomycin). The investigators hypothesize that there will be no difference in complication (infection) rates between groups.

ELIGIBILITY:
Inclusion Criteria

* Patient is undergoing total ankle arthroplasty.
* Patient is able to give informed consent to participate in the study. LAR consents will not be utilized for this study
* Age Range >18

Exclusion Criteria

* Previous lower extremity surgery that in the opinion of the principal investigator or qualified research personnel precludes the participant from safely participating on the study.
* BMI > 40.
* Contraindication to receiving vancomycin, cefepime, ancef, or other standard of care pre-operative antibiotic (allergy, medical issue, etc).
* Inability to administer the IO infusion.
* Patient refusal to participate.
* Uncontrolled Diabetes Mellitus type 1 or 2, defined as Hemoglobin A1C >7.5.
* Immunocompromised or immunosuppressed patients (HIV, Hep C, end stage renal disease, dialysis, transplant, chemo/radiation treatment in last 6 months, medications).
* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Systemic Sample Vancomycin Tissue Concentration - Start of Case | perioperatively
Systemic Sample Vancomycin Tissue Concentration - End of Case | perioperatively
Capsule or Synovium Sample Vancomycin Tissue Concentration | immediately after the procedure
Distal Tibia Sample Vancomycin Tissue Concentration | immediately after the procedure
Talar Bone Sample Vancomycin Tissue Concentration | immediately after the procedure

SECONDARY OUTCOMES:
90 day post-operative wound complication and infection rates | 90 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Ahuero, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided